CLINICAL TRIAL: NCT05818514
Title: A Phase 0 Open Label Positron Emission Tomography Study to Assess the Biodistribution and Binding Characteristics of [11C]AZ14132516 Following Administration to Healthy Participants
Brief Title: A PET Study to Determine Biodistribution and Binding Characteristics of [11C]AZ14132516 in Healthy Participants
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: D9690C00003
Record Dates: First submitted 2023-03-15; First posted 2023-04-19 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [11C]AZ14132516 (Experimental): Pilot panel: up to 3 participants to complete 1 PET examination each during the course of the study Main panel: up to 6 participants to complete 2 PET examinations each during the course of the study
  Interventions: Drug: [11C]AZ14132516

INTERVENTIONS:
Drug: [11C]AZ14132516 — Injection of radioligand for PET examinations
  Other Names: No other names

SUMMARY:
The purpose of this study is to measure the regional distribution and binding of [11C]AZ14132516 to CCR9 in the abdomen using PET-CT examination in healthy participants.

Study details include:

The study duration will be up to 60 days.

The IV radioligand [11C]AZ14132516 will be administered at PET-CT examination: Visit 2 for the pilot panel; Visit 2 and 3 in the main panel.

There will be 2 study visits for the pilot panel and 3 study visits for the main panel.

DETAILED DESCRIPTION:
This is a Phase 0, first in human (FIH) open label radioligand development study in healthy male and female participants. This radioligand development study will consist of two sequential panels:

Pilot panel (n = up to 3) Main panel (n = up to 6)

The purpose of the pilot panel is to perform initial PET-CT examinations using radioligand [11C]AZ14132516 and to optimise the imaging protocol. Up to 3 participants are planned to be included in this panel. Participants will attend the PET unit for a single visit and will be administered a single intravenous microdose of [11C]AZ14132516 (≤ 10μg regardless of body weight, approximately 400 MBq/70kg radioactivity) followed by a single PET-CT examination.

The purpose of the main panel is to assess [11C]AZ14132516 kinetics, binding characteristics, develop the quantitative analysis protocol and assess reproducibility of the analysis. Six participants are planned to be included in this panel. Participants will attend the PET unit for a baseline visit with administration of a single intravenous microdose of [11C]AZ14132516 followed by a PET-CT examination. Participants will return for a repeat visit 10 to14 days later where a second intravenous microdose of [11C]AZ14132516 will be administered followed by a second PET-CT examination.

ELIGIBILITY:
Inclusion Criteria:

Informed Consent

1. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in the protocol.
2. Able and willing to participate in all scheduled evaluations, abide by all study restrictions, and complete all required tests and procedures.
3. Participants ≥ 20 to 65 years of age inclusive, at the time of signing the ICF.
4. Participants who are healthy as determined by medical evaluation including medical history, physical examination, laboratory parameters and ECG performed before first administration of investigational product.
5. Body weight within 50.0 to 100.0 kg and body mass index within the range 18.0 to 30.0 kg/m2 (inclusive).
6. Contraceptive use by males or females should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

   1. Female participants:

      In this study:
      * WOCBP must have a negative pregnancy test at screening and before PET examination (all premenopausal women, or in case when menstrual status cannot be ascertained in women under the age of 55 years).
      * If sexually active with a non-sterilised male partner, must use at least one highly effective method of birth control during the study period and for 7 days following last radioligand administration.

      It is strongly recommended that non-sterilised male partners of female participants of childbearing potential use a male condom plus spermicide during the study period.

      Female participants must not breastfeed and must not donate or retrieve ova for their own use during the study period and for 7 days following last radioligand administration.
   2. Male participants:

      * Non-sterilised male participants who are sexually active with a female partner of childbearing potential must use a condom with spermicide during the study period and for 7 days following last radioligand administration. It is strongly recommended that female partners of male participants also use at least one highly effective method of contraception throughout this period. In addition, male participants must refrain from fathering a child or donating sperm during the study period and for 7 days following last radioligand administration.

Exclusion Criteria:

1. Current significant major or unstable respiratory disease, heart disease, cerebrovascular disease, hematological disease, hepatic disease, renal disease, gastrointestinal disease, or other major diseases.
2. Participants with unstable hypertension (as judged by the Investigator) or symptomatic hypotension, history of pre-syncope or syncope due to orthostatic hypotension and/or induced by change of posture (orthostatic hypotension defined as 25 mmHg decrease in systolic and/or 15 mmHg).
3. Significant abnormalities on the clinical examination, including neurological and physical examination, vital signs, ECG and clinical.
4. Chemistry, hematology, or urine analysis results that may interfere with the study or present a safety risk to the patient.
5. Abnormal vital signs, after 10 minutes of supine rest as judged by the PET centre physician. As a guide, any readings outside the following should be considered in the evaluation:

   1. systolic blood pressure (BP) ≥ 140 mmHg
   2. diastolic BP ≥ 90 mmHg
   3. heart rate ≤ 35 bpm or ≥ 100 bpm The inclusion of participants meeting the above criteria may be decided on a case-by case basis by PET centre physician.
6. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG that may interfere with the interpretation of QTc interval changes. This may include participants with any of the following:

   1. PR (PQ) interval prolongation of clinical significance as judged by the Investigator
   2. Intermittent second or third degree AV block (AV block II Mobitz type 1, Wenchebach, while asleep or in deep rest is not disqualifying)
   3. Incomplete, full, or intermittent bundle branch block (QRS ≤ 110 ms with normal QRS and T wave morphology is acceptable if there is no evidence of left ventricular hypertrophy)
   4. Abnormal T wave morphology, particularly in the protocol-defined primary lead
   5. Prolonged QTcF ≥ 470 ms or shortened QTcF ≤ 340 ms or a family history of long QT syndrome.

   The inclusion of participants meeting the above criteria may be decided on a case-by case basis by PET centre physician.
7. Known or suspected systemic infection (eg, hepatitis B virus, hepatitis C virus, HIV and tuberculosis), including previous or ongoing infectious or autoimmune disease.
8. Participants must abstain from taking prescription or non-prescription drugs (including vitamins, recreational drugs, and dietary or herbal supplements) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) before the start of study intervention until completion of the follow-up visit, unless, in the opinion of the investigator and sponsor, the medication will not interfere with the study.
9. Current drug abuse or dependence or positive screen for drugs of abuse at screening visit.
10. Participants on anticoagulant treatment.
11. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
12. Suffers from claustrophobia that limits the ability to undergo the scanning procedure.
13. Participant has abnormal blood flow confirmed by a negative Allen's test in both hands at screening.
14. Blood donation within 1 month of screening or any blood donation/blood loss greater than 500 mL during the 3 months prior to screening.
15. Positive SARS-CoV-2 rapid antigen test at screening
16. Any other reason that, in the study PI opinion, prohibits the inclusion of the participants into the study.
17. Judgement by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.

    -

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2023-07-11 (Actual)

PRIMARY OUTCOMES:
SUV and SUVR in abdominal regions of interest | Immediately following administration of radioligand
  Standardized uptake value (SUV) is the radioactivity concentration in given region of interest normalized for injected radioactivity and body weight.
  Standardised uptake value ratio (SUVR) is the ratio of SUV in a given region of interest to a reference region without significant radioligand uptake

SECONDARY OUTCOMES:
Absolute percentage differences of SUV and SUVR, and intraclass correlation coefficients, in regions of interest between two test-retest PET examinations | 10-14 days following initial administration of radioligand
Number of participants with safety findings, AEs | Through study completion, up to 49 days (including screening period)

OTHER OUTCOMES:
Quantitative estimates of total and specific binding (Kp, VT), including cross-validation of different image analysis approaches | Immediately following administration of radioligand

CONTACTS AND LOCATIONS:
Overall Officials: Per Stenkrona, Principal Investigator — Karolinska Institutet
Locations (1):
- Research Site, Solna, Sweden